CLINICAL TRIAL: NCT06045182
Title: Additional Effects of Piriformis Stretch in the Management of Sacroiliac Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/16
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Sacroiliac Joint
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive maitland mobalizations and the second will receive maitland mobalization along with piriformis stretch. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Maitland mobalizations ) (Active Comparator): Patients in this group will receive Maitland mobilizations along with hot pack and TENS for pain and disability. A total of 3 sessions would be conducted over a period of 1 week.
  Interventions: Procedure: Maitland mobilization; Procedure: Electrotherapy
- Group B (Maitland Moblizations along with piriformis stretch) (Experimental): Patients will receive Maitland mobilizations along with hot pack and TENs and additional stretch of piriformis muscle is given. A total of 3 sessions would be conducted over a period of 1 week.
  Interventions: Procedure: Maitland mobilization; Procedure: Piriformis stretch; Procedure: Electrotherapy

INTERVENTIONS:
Procedure: Maitland mobilization — Participants in this group will be first given hot pack and TENS for 10 min. Then they will be given Maitland Mobilizations (10 oscillations total of 3 sets )with 10 sec rest in between. Mobilization will be Unilateral or central based on the patient condition and Intensity of Mobilizations increases as per patient tolerance in 2nd and 3rd session.
Procedure: Piriformis stretch — Piriformis stretch will be given to this group. In first session piriformis stretch will be given for 10 sec with 10-second resting time in between with, 7 rep total of 1 set. For the 2nd and 3rd session repetitions will be increase to 8 and 10 respectively.
  Arms: Group B (Maitland Moblizations along with piriformis stretch)
Procedure: Electrotherapy — Hot pack and TENS for 10 min

SUMMARY:
Sacroiliac joint (SIJ) dysfunction is known as an important contributing factor in lower back pain. Pain and stiffness experienced from the sacroiliac joint in the SI region (hips/groins or may spread to lower extremity) is referred as SIJ dysfunction.Physiotherapists have a wide range of options in managing SIJD including Manipulation, Kinesiotaping, Muscle Energy Technique (MET), McKenzie, Maitland's mobilization, and Mulligan's mobilization. So far studies have shown the efficacy of different treatment tools in combination or in isolation. Likewise, researchers have also studied the effect of piriformis stretch in combination with other exercises on sacroiliac joint pain. However, there is very limited literature available on the cumulative effect of piriformis stretch along with mobilization maneuvers on pain and disability in patient with SIJ dysfunction.Since piriformis is one of the most important muscles involved in stabilization of SI joint and a major source of SI dysfunction, hence the current study is designed to investigate the additional effects of piriformis stretch with manual therapy in the management of sacroiliac joint dysfunction.

DETAILED DESCRIPTION:
SIJ dysfunction is a prominent source of pain in low back pain patients. It is reported that 10-30% of individuals suffering from lower back pain is due to SIJ dysfunction.There are different risk factors for developing SIJ dysfunction including leg length discrepancies, a history of lumbar fusion, scoliosis, sustained athletic activity, pregnancy, spondyloarthropathies, or gait abnormalities.Muscles that are commonly found to be shortened (or tightened) in SIJ dysfunction include the rectus femoris, tensor fascia Lata, hip adductors, quadratus lumborum, piriformis, obturator internus, and latissimus dorsi. Particular attentions should be directed to the piriformis muscle. t alters the SIJ motion by rotating the sacrum to the opposite side.Continued inflexibility of this muscle is often thought to be part of the source of recurrent pain Over time several treatment aporaches have been developd to treat SIJ dysfunction.Clinicians also use different electrotherapy modalities, biomechanical correction techniques, and exercises for addressing SI joint pain. Many therapeutic exercises including piriformis stretch, muscle activation exercises and exercise therapy have the potential of improving sacroiliac joint dysfunction , however evidence is deficient. This research presents additional effects of piriformis stretch in the management of sacroiliac joint dysfunction.It will expand current understanding of effects of piriformis stretch on disability and pain in patients with SIJ dysfunction and help in providig treatment protocols for improving pain in patients with sacroiliac joint dysfunction.

Main objective of thi study is to determine and compare the effect of piriformis stretch along with mobilization as compared to SIJ mobilization alone on pain and disability in patients with SIJ dysfunction.

The participants meeting the eligibility citeria will be recruited, followed by random allocation to 2 groups. Both groups will recive standard treatment protocol which consists of Hot pack TENs, mobalization.Three sessions will be provided on alternative days. Pre and Post assessment of pain and disability will be noted

ELIGIBILITY:
Inclusion Criteria:

* Adults (both male and female) aged 18-45 years experiencing sacroiliac joint pain
* Patients fulfilling the diagnostic criteria, recommended by the International Association for the Study of Pain (IASP).(13)
* Those with > 4 score on Numeric pain rating scale for the sacroiliac pain
* Using no other pain killers or non steroidal anti-inflammatory drugs during the therapy

Exclusion Criteria:

* Individuals suffering from pain due to other conditions (low back pain, hip pathology, hip osteoarthritis, cognitive disorders, radicular pain, ankylosing spondylitis, coccydynia)
* Patients with piriformis syndrome.
* SIJ pain due to other causes such as fractures, tumors and trauma.
* Pregnant females
* Those patients who have received any surgical treatment for SIJ dysfunction

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 1 week
  Pain will be measured using the Numeric Pain Rating Scale, which is an 11-item scale
Disability level of participant | 1 week
  Disability will be assessed using Oswestry low back disability Index. A higher score indicates more disability

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan